CLINICAL TRIAL: NCT05974475
Title: MONDRIAN: Multi-omics Integrative Modelling for Stereotactic Body Radiotherapy in Early-stage Non-small Cell Lung Cancer
Acronym: MONDRIAN
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Sponsor
Other Study IDs: R1842/23-IEO1973
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Lung Neoplasm Malignant
Keywords: Early stage non-small cell lung cancer; Stereotactic body radiotherapy (SBRT); Radiosensitivity; Radioresistance; Multi-omics; Radiomics; Genomics; Proteomics; Outcome modeling
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiosurgery; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Formalin-fixed paraffin-embedded (FFPE) bioptic samples (SBRT cohort); formalin-fixed paraffin-embedded (FFPE) surgical specimens (surgical cohort)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SBRT Cohort: Radiation: Stereotactic Body Radiotherapy (SBRT)
  Interventions: Radiation: SBRT
- Surgery Cohort: Procedure: Surgery
  Interventions: Procedure: Surgery

INTERVENTIONS:
Radiation: SBRT — State-of-art SBRT will be delivered in 3-5 fractions; prescription doses and fractionation schedules will be defined according to patient- and tumor-related characteristics (e.g. pulmonary comorbidities, tumor location: peripheral vs central vs ultra-central).
  Other Names: Stereotactic body radiotherapy; Stereotactic Ablative Radiotherapy (SABR)
  Groups: SBRT Cohort
Procedure: Surgery — State-of-art surgery will be consist in pulmonary anatomical resection (i.e. segmentectomy or lobectomy) and systematic lymph node dissection.
  Groups: Surgery Cohort

SUMMARY:
Stereotactic Body Radiotherapy (SBRT) is a form of high-precision radiotherapy playing a major role in patients diagnosed with early-stage non-small cell lung cancer (NSLCL), especially when surgery cannot be performed. It is a non-invasive, well-tolerated treatment, with an excellent ability to control disease recurrence. However, in some patients, disease response is suboptimal: understanding why this happens may open doors to more aggressive approaches, such as the combination with systemic therapies.

Hence, the goal of this observational trial is to understand which clinical, imaging, and biological factors are associated with response to SBRT through the development of complex models. In other words, the main question it aims to answer is: "Will this patient respond to radiation treatment based on the characteristics of their disease?".

Participants will be treated according to the best clinical practice standards, in agreement with international, national, and internal guidelines.

Researchers will compare data collected from patients treated with SBRT with those collected from a similar group of patients, who will be treated with surgery, to see which factors are actual predictors of response to SBRT, or rather are indicators of more or less aggressive disease behavior.

DETAILED DESCRIPTION:
The overall planned duration of the study is 60 months.

The project is structured into five main tasks, as following:

* Task 1_Clinical study: Routine clinical data will be collected from eligible patients, including demographics, disease and treatment characteristics, pulmonary function, and blood count parameters.
* Task 2_Radiomics study: Quantitative imaging analysis will be performed on both diagnostic computed tomographies (CTs) and positron emission tomographies (PETs). A software compliant with the Imaging Biomarker Standardization Initiative (IBSI) will be used to extract radiomic features at baseline and at the first clinical progression (or at the last available follow-up, whichever comes first). Clinically established qualitative and semiquantitative metrics (e.g. pleural effusion in CT images and standardized uptake value in PET images) will be retrieved, as well.
* Task 3_Gene expression study: Gene expression profiling will be performed at baseline in both cohorts to investigate the presence of a prognostic pretreatment signature. The analysis will be performed on formalin-fixed paraffin-embedded (FFPE) tissue samples (namely, resected tumor in the surgical cohort and bioptic sample- whenever available- in the SBRT group). A next-generation sequencing (NGS)-based assay which targets 395 immune-related genes and named as Oncomine™ Immune Response Research Assay, will be employed.
* Task 4_Proteomics study: Proteomics will integrate the study of RNA expression performed in Task 3. As in Task 3, the analysis will be performed on FFPE samples, from both patients' cohorts.
* Task 5_Integrative model building: Integration of all previous features in a unique classification model able to determine a precise estimate of individuals with high vs low risk of disease progression and, at the same time, identify relevant predictive factors. The proposed classification model will integrate data from different sources using a multi-layer deep neural network. Federated learning techniques will also be used to reduce the bias due to the choice of a specific trial or data source.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven NSCLC; all histologies will be considered eligible (e.g. squamous, adenocarcinoma, large cell carcinoma);
* American Joint Committee on Cancer Tumor Node Metastasis (AJCC TNM) classification (8th Edition) clinical stage I-II;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
* No absolute contraindications to either surgery (e.g. severe comorbidities) or SBRT (e.g. active connective diseases, severe pulmonary fibrosis);
* Ability and willingness to sign a written informed consent for treatment and study participation.

Exclusion Criteria:

* Prior diagnosis of invasive cancer (within 3 years before the diagnosis of ES-NSCLC);
* Mental diseases or psychiatric disorders preventing the acquisition of a valid informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care cancer center, early-stage NSCLC.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 24 months
  The time between the beginning of SBRT or date of surgery, and any disease progression (local, regional, distant), death from any cause, or last follow-up, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Volpe, MD, Principal Investigator — Istituto Europeo di Oncologia IRCCS
Locations (2):
- Italy (2):
  - Istituto Europeo di Oncologia IRCCS, Milan, Italy
  - Istituto Europeo di Oncologia (IEO) IRCCS, Milan, Lombardy

REFERENCES:
- [Derived] Volpe S, Zaffaroni M, Piperno G, Vincini MG, Zerella MA, Mastroleo F, Cattani F, Fodor CI, Bellerba F, Bonaldi T, Bonizzi G, Ceci F, Cremonesi M, Fusco N, Gandini S, Garibaldi C, Torre D, Noberini R, Petralia G, Spaggiari L, Venetis K, Orecchia R, Casiraghi M, Jereczek-Fossa BA. Multi-omics integrative modelling for stereotactic body radiotherapy in early-stage non-small cell lung cancer: clinical trial protocol of the MONDRIAN study. BMC Cancer. 2023 Dec 15;23(1):1236. doi: 10.1186/s12885-023-11701-9. PMID 38102575